CLINICAL TRIAL: NCT02381067
Title: A Prospective, Efficacy Study of NuCel® in Patients Undergoing Fusion for One, Two or Three Level Degenerative Disease of the Cervical Spine
Brief Title: A Prospective Study of NuCel® in Cervical Spine Fusion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure of PI from the study facility
Sponsor: NuTech Medical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD2015-01-01
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Spondylosis; Spinal Stenosis; Spondylolisthesis; Intervertebral Disc Disease; Intervertebral Disc Degeneration
Keywords: Cervical Fusion; NuCel; Amniotic Allograft; Prospective
MeSH Terms: conditions — Spondylosis; Spinal Stenosis; Spondylolisthesis; Intervertebral disc disease; Intervertebral Disc Degeneration; Klippel-Feil Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NuCel with Allograft Bone (Other): NuCel will be used with allograft bone for the surgical treatment of one, two or three level degenerative disease of the cervical spine.
  Interventions: Other: NuCel with Allograft Bone

INTERVENTIONS:
Other: NuCel with Allograft Bone — NuCel is a minimally manipulated allograft product derived from amniotic membrane along with cells from amniotic fluid. Allograft bone is bone that comes another patient. NuCel and Allograft bone will be combined for this treatment.

SUMMARY:
The study is intended to demonstrate that the NuCel® allograft is effective and safe in promoting bone growth and fusion rate when used in cervical fusion in patients with one, two or three-level diseases of the cervical spine.

DETAILED DESCRIPTION:
The study is intended to demonstrate that the NuCel® allograft is effective and safe in promoting bone growth and fusion rate when used in cervical fusion in patients with one, two or three-level diseases of the cervical spine. Sixty subjects will participate in the study at a single clinical site. Participants will be at least 21 years of age. All subjects will have been established with cervical spine disease at one, two or three levels of the cervical spine that requires cervical interbody fusion per the opinion of the treating surgeon. The primary objective is to demonstrate that NuCel® is comparable to autograft bone graft in producing a successful, contiguous fusion at 6 months ±4 weeks post-operative when used in cervical fusion surgery. Success based on findings of cervical CT scan and plain radiographs. Additionally, Visual Analog Scale (VAS), Neck Disability Index (NDI) and patient satisfaction will be used as secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 21 years of age
2. Have clinical and radiological evidence of degenerative disc disease, spondylosis, spinal stenosis, or spondylolisthesis at either one, two or three levels of cervical spine.
3. In the opinion of the treating surgeon, must already be a qualified candidate for cervical fusion surgery.
4. Be likely to return for regular follow-ups until the end of the study period.
5. Be willing and able to provide Informed Consent for study participation.

Exclusion Criteria:

1. Neck pain due to acute trauma.
2. Clinical, laboratory and/or radiological evidence of neck pain secondary to acute or chronic infection, malignancy, other space occupying lesions and metabolic bone demineralization diseases (e.g. osteomalacia, gout, Paget's disease etc.).
3. Any terminal or autoimmune disease including but not limited to HIV infection, or rheumatoid arthritis.
4. Any other concurrent medical disease or treatment that might significantly impair normal healing process as evaluated by the PI.
5. Recent history (within past 6 months) of any chemical or alcohol dependence requiring treatment.
6. Currently a prisoner.
7. Currently experiencing a major mental illness (psychosis, schizophrenia, major affective disorder) which may indicate that the symptoms are psychological rather than of physical origin.
8. Pregnancy at the time of enrollment.
9. In order to confirm eligibility, subjects previously diagnosed with osteoporosis, osteopenia or osteomalacia, female subjects over the age of 65, post-menopausal female subjects under the age of 65 with any of the risk factors for osteoporosis, and subjects at the investigator's discretion will have DEXA scans performed prior to study entry. If DEXA is required, exclusion will be defined as a DEXA bone density measurement T score ≤ -2.5

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Interbody Fusion measured using CT scans and standard radiographs | 6 months
  Interbody fusion will be measured using CT scans and standard radiographs

SECONDARY OUTCOMES:
Change from baseline pain using Visual Analogue Scale (VAS) | 6 weeks, 3 months, 6 months, 1 year
Change from baseline Neck Disability Index (NDI) | 6 weeks, 3 months, 6 months, 1 year
Patient Satisfaction Survey | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Franklin Lin, M.D., Principal Investigator — Wellstar Hospital
Locations (1):
- Wellstar Hospital, Marietta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No